CLINICAL TRIAL: NCT07036900
Title: Effects of Flexion and Extension Type Arm Slings on Walking Kinematics and Balance in Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Ceren Bayrak (Other)
Responsible Party: Sponsor-Investigator, Ceren Bayrak, PhD (c), Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Other Study IDs: ODGQzpAt
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Arm Slings; Walking Kinematics; Balance; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients (experimental group (EG)): All test assesments were explained to the patient both verbally and visually. All assesments were applied for patients and healthy participants on the same day. Patients using assistive devices were assessed with these devices. Participants were initially assessed for gait analysis without an arm sling. Then, assessments were conducted by applying a flexor arm sling first, followed by an extensor arm sling. The assessments and data collection were conducted by physiotherapists.
- Healthy individuals (control group (CG)): All test assesments were explained to the patient both verbally and visually. All assesments were applied for patients and healthy participants on the same day. Patients using assistive devices were assessed with these devices. Participants were initially assessed for gait analysis without an arm sling. Then, assessments were conducted by applying a flexor arm sling first, followed by an extensor arm sling. The assessments and data collection were conducted by physiotherapists.

SUMMARY:
In the clinic, stroke patients are seen to use flexor or extensor type arm slings, but no study was found investigating the effects of these different types of arm slings on walking kinematics and balance. The aim of the presented study was to investigate the effects of different types of arm slings on walking kinematics and balance in stroke patients and to compare them with healthy individuals.

DETAILED DESCRIPTION:
Stroke is one of the most common diseases in the world, affecting one in every four people (Campbell & Khatri, 2020). After stroke, approximately 80% of patients experience walking disorders (Algurén et al., 2010). Stroke survivors demonstrate gait disturbances such as reduced walking speed, step length and cadence (Balaban & Tok, 2014). Deterioration in walking kinematics negatively affects daily living activities, confidence, self-care, social roles, family life and reducing quality of life in stroke survivors (Park & Kim, 2019). Additionally, walking disturbances in stoke patients can lead to increased energy expenditure, pain and risk of falling (Balaban & Tok, 2014; Shin et al., 2020). Besides, balance impairments are frequent clinical symptom in stroke survivors. Compared to healthy individuals, stroke patients have lower balance and walking capacity. Accordingly, the risk of falling increases, physical activity and participation reduces in individuals with stroke (Roelofs et al., 2023). Therefore, it is important that walking kinematics and balance in stroke survivors should have similar characteristics to the healthy individuals.

One of the frequently complications after stroke is shoulder subluxations. Shoulder subluxation increases the distance between the acromion and the humeral head, thus delay improvement of upper extremity motor function and decrease proprioception in stroke survivors (Paci et al., 2005). Electrical stimulation, robot-assisted upper extremity rehabilitation and arm slings are the physiotherapy and rehabilitation applications used to prevent shoulder subluxations in stroke patients (Jung & Choi, 2019; Paci et al., 2005). Arm slings are often used to help reposition the humeral head in the glenoid fossa by counteracting gravity on the affected side (Jeong et al., 2022). In addition, it has been stated that arm slings have a positive effect on balance, increase walking efficiency, reduce spasticity and are a painless application in stroke survivors (Acar & Karatas, 2010; Jeong et al., 2022). In the clinic, it has been observed that stroke patients use flexor or extensor type arm slings. However, no study has been found investigating the effects of these different types of arm slings on walking kinematics and balance in stroke patients. The aim of the presented study is to investigate different types of arm slings on walking kinematics and balance in stroke patients and compare with the healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for EG were: (1) stroke diagnosis, (2) age 18-80, (3) independent ambulation (Functional Ambulation Category-FAS ≥ 2), (4) Modified Ashworth Scale-MAS ≤2 for gastrocnemius and biceps muscles, (5) ability to walk 10 m independently or with assistive device, (6) physician approval for an exercise program.
* Inclusion criteria for CG: (1) healthy individuals without any additional neurological or orthopaedic diseases that may affect balance and gait, (2) age 18-80, (3) physician approval for an exercise program.

Exclusion Criteria:

* (1) severe visual impairments, (2) cerebellar involvement, (3) upper extremity Brunnstrom stage ≤ 3, (4) cancer diagnosis, (5) presence of a neurological or orthopedic condition other than stroke, (6) inability to understand and follow commands or lack of cooperation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective, randomized controlled study involved ambulatory stroke patients (experimental group (EG)) and healthy individuals (control group (CG)).
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
PABLO ® Lower Extremity inertial sensor | 8 min.
  Inertial measurement unit (IMU) systems have been validated for measuring joint angles and temporal characteristics during lower extremity movements (O'Reilly et al., 2018). Gait parameters, such as stance and swing phase durations, step length, walking speed, and cadence, can be determined using two inertial sensors placed in the shoes. Each shoe is equipped with a PABLO Lower Extremity Inertial Sensor. The sensors measure angular velocity and acceleration at a sampling frequency of 110Hz. Each sensor transmits data via Bluetooth. The sensors are attached to the participants' shoes using custom Velcro straps. It has been found that inertial measurement unit systems work reliably not only in healthy individuals but also in patients, providing accurate results under different pathological gait patterns (Laidig et al., 2021). In our study, gait analysis was conducted to establish reference values by evaluating stroke patients and healthy individuals of the same age.
TYMO ® Balance Plate | 8-10 min.
  The TYMO® Balance Plate (Tyromotion, Austria) is a standardized balance analysis device used to assess posture and balance in an upright stance. The TYMO® force sensors detect weight shifting and measure the center of pressure, body sway, and load balance on the feet. These data provide indicators of balance, stability, and symmetry. The TYMO® system is a versatile and easy-to-use assessment and treatment tool consisting of the TYMO Therapy Board and software. Participants are required to stand on a platform for 30 seconds and undergo four test positions: 1) feet apart, eyes open, firm support surface; 2) feet apart, eyes closed, firm support surface; 3) feet apart, eyes open, soft support surface/foam; 4) feet apart, eyes closed, soft support surface/foam. Each position was tested once, and the displacement of the center of body mass was measured in centimeters (Dudoniene et al., 2023).

SECONDARY OUTCOMES:
Timed Up and Go Test | 3-5 min.
  The Timed Up and Go test is used to assess a person's walking speed, fall risk, and mobility (Wall et al., 2000). In this test, the patient is instructed to stand up from a chair, walk a previously marked 3-meter distance, turn, and then return to sit back down in the chair. The average time in seconds is recorded after three repetitions to find the result. A completion time longer than 13.5 seconds is considered indicative of an increased fall risk, while a time exceeding 20 seconds is associated with decreased mobility (Podsiadlo & Richardson, 1991).

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçeşehir Liv Hospital Neur-on, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned that patient data will not be shared with anyone.

REFERENCES:
- See also: article — https://doi.org/10.1016/j.gaitpost.2010.09.008
- See also: article — https://doi.org/https://doi.org/10.1016/S0140-6736(20)31179-X
- See also: article — https://doi.org/10.12965/jer.1734898.449
- See also: article — https://doi.org/10.3389/fdgth.2021.736418
- See also: article — https://doi.org/10.1038/s41598-021-90602-y
- See also: article — https://doi.org/10.1007/s40279-018-0878-4